CLINICAL TRIAL: NCT06972485
Title: Comparison of Hemodynamic Effects of Hypobaric and Hyperbaric Bupivacaine in Spinal Anesthesia During Hip Surgery in Geriatric Patients
Brief Title: Comparison of Hemodynamic Effects of Hypobaric and Hyperbaric Bupivacaine in Spinal Anesthesia in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Fadime Alagaş, Research assistant, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FALAGAS 1
Record Dates: First submitted 2025-04-30; First posted 2025-05-15 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-04

CONDITIONS: Geriatric Patient; Spinal Anesthesia; Hip Surgery
Keywords: Geriatric patient; Hemodynamic changes; Hypobaric bupivacaine; hyperbaric bupivacaine
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Intervention will be performed in geriatric patients of hemodynamic changes (hypotension, bradycardia) associated with spinal anesthesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HypoB (Active Comparator): In the HypoB group, spinal anesthesia will be administered intrathecally using 3 cc of hypobaric bupivacaine solution in the lateral decubitus position, with the fractured side positioned upward.The patients will then be kept in the lateral position for 15 minutes. The patients' hemodynamic data , bilateral sensory and motor block levels will be recorded.
  Interventions: Procedure: spinal anesthesia
- HyperB (Active Comparator): In the HyperB group, spinal anesthesia will be administered intrathecally using 3 cc of hyperbaric bupivacaine solution in the lateral decubitus position, with the fractured side positioned downward.The patients will then be kept in the lateral position for 15 minutes. The patients' hemodynamic data, bilateral sensory, and motor block levels will be recorded.
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — spinal anesthesia with hypobaric and hyperbaric bupivacaine

SUMMARY:
The frequency of hypotension is increased in geriatric patients due to physiological changes compared to the normal population. In this study, our aim is to compare the hemodynamic changes in geriatric patients undergoing hip surgery under spinal anesthesia with hypobaric and hyperbaric bupivacaine.

DETAILED DESCRIPTION:
Patients will be randomly assigned to one of two groups: HypoB (% 0.5 bupivacaine 3cc+ 2cc distilled water) or HyperB (% 0.5 bupivacaine 3cc+ 2cc %10 dextrose). For pre-positioning analgesia, an intravenous dose of fentanyl at 0.5 mcg/kg will be administered. Patients will then be positioned in the appropriate lateral decubitus position based on whether hypobaric or hyperbaric bupivacaine is used. Spinal anesthesia will be performed using 3 cc local anesthetic solution, followed by 15 minutes of lateralization.

During the surgery, hemodynamic parameters, sensory block levels at the 5th, 10th, 15th, and 20th minutes at lateral and supine position, and motor block levels with bromage scale at the 15th and 20th minutes at supine position will be recorded. The spread of the block to the T8 dermatome level was considered an indicator of a successful block. Hemodynamic parameters (blood pressure, heart rate, peripheral oxygen saturation) will be recorded at 0, 5, 10, 15, 20, 30, 40, 50, 60, 90, and 120 minutes intraoperatively. Patients will receive crystalloid infusion at a rate of 5-7 ml/kg per hour throughout the procedure. The volume of intraoperative bleeding, the amount of blood products administered, and the doses of ephedrine, atropine, and noradrenaline used will also be documented. If the heart rate falls below 45 beats per minute, 0.5 mg of intravenous atropine will be administered.

A decrease in blood pressure of 20% or more from baseline will be defined as hypotension. In such cases, ephedrine will be administered. If hypotension persists despite a total dose of 20 mg ephedrine, a noradrenaline infusion will be initiated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age
* Patients taken to surgery in a supine position due to femur fractures
* Patients classified as ASA (American Society of Anesthesiologists) class I-III

Exclusion Criteria:

* History of allergy to the drug
* Patients with coagulopathy
* Patients refusing to participate in the study
* Severe valve stenosis
* Infection at the injection site
* Inadequate spinal anesthesia level during surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-27 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Hemodynamic effects of hypobaric and hyperbaric bupivacaine with spinal anesthesia | 2 hour
  blood pressure monitoring

SECONDARY OUTCOMES:
Evaluation of sensorial block with hypobaric and hyperbaric bupivacaine in spinal anesthesia | 2 hour
  sensorial block evaluate with pinprick test; sensorial block level; present/absent
Evaluation of motor block with hypobaric and hyperbaric bupivacaine in spinal anesthesia | 2 hour
  motor block evaluate with bromage scale ;Grade 0: Full movement of hips, knees, and ankles (no block). Grade 1: Unable to lift the leg but can move knees and ankles (partial block). Grade 2: Unable to bend the knee but can move ankles (near-complete block). Grade 3: No movement in hips, knees, or ankles (complete block).

CONTACTS AND LOCATIONS:
Overall Officials: Sacit Güleç, Professor, Study Director — Eskisehir Osmangazi University
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Odunpazari, Turkey (Türkiye)

REFERENCES:
- [Background] Herrera R, De Andres J, Estan L, Olivas FJ, Martinez-Mir I, Steinfeldt T. Hemodynamic impact of isobaric levobupivacaine versus hyperbaric bupivacaine for subarachnoid anesthesia in patients aged 65 and older undergoing hip surgery. BMC Anesthesiol. 2014 Oct 24;14:97. doi: 10.1186/1471-2253-14-97. eCollection 2014. PMID 25371654
- [Background] Uppal V, Retter S, Shanthanna H, Prabhakar C, McKeen DM. Hyperbaric Versus Isobaric Bupivacaine for Spinal Anesthesia: Systematic Review and Meta-analysis for Adult Patients Undergoing Noncesarean Delivery Surgery. Anesth Analg. 2017 Nov;125(5):1627-1637. doi: 10.1213/ANE.0000000000002254. PMID 28708665
- [Background] Gong C, Ye X, Liao Y, Ye P, Zheng T, Zheng X. Hypotension after unilateral versus bilateral spinal anaesthesia: A Systematic review with meta-analysis. Eur J Anaesthesiol. 2025 Mar 1;42(3):203-223. doi: 10.1097/EJA.0000000000002098. Epub 2024 Nov 21. PMID 39575900